CLINICAL TRIAL: NCT01513044
Title: An Open-label, Balanced, Randomized, Two-treatment, Two-period, Two Sequence, Single Dose, Crossover, Bioequivalence Study in Healthy, Adult,Human, Male Subjects Under Fasting Conditions.
Brief Title: Bioequivalence Study of Mycophenolate Mofetil 250 mg Capsule, Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 08-VIN-182
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: bioequivalence; Mycophenolate Mofetil; crossover
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mycophenolate Mofetil (Experimental): Mycophenolate Mofetil 250 mg capsules of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Mycophenolate Mofetil
- Cellcept (Active Comparator): Cellcept 250 mg capsules of Roche Laboratories Inc.
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Mycophenolate Mofetil 250 mg capsules of Dr. Reddy's Laboratories Limited
  Arms: Mycophenolate Mofetil
Drug: Mycophenolate Mofetil — 250 mg capsules of Roche Laboratories Inc.
  Other Names: Cellcept
  Arms: Cellcept

SUMMARY:
An open-label, balanced, randomized, two-treatment, two-period, two sequence, single dose, crossover, bioequivalence study of Mycophenolate mofetil 250 mg Capsule of Dr. Reddy's Laboratories limited, comparing with that of Cellcept 250 mg Capsule of Roche Laboratories in healthy, adult,human, male subjects under fasting conditions.

DETAILED DESCRIPTION:
This was an open-label, balanced, randomized, two-treatment, two-sequence, two-period, single dose, crossover bioequivalence study in healthy, adult, human, male subjects under Fasting conditions. 72 healthy male adults were enrolled. A washout period of 7 days was maintained between the successive dosing days.One capsule containing mycophenolate mofetil 250 mg was administered orally with 240 mL water in sitting posture, after an overnight fast of at least 10 hours in each period. This activity was followed by a mouth check to assess compliance to dosing. The subjects were not allowed to lie down for the first two hours after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 50 years (including both).
* Subjects' weight within the normal range according to normal values for the Body
* Mass Index (1 8.5 to 24.9 kg/m2) with minimum of 50 kg weight.
* Subjects with clinically acceptable normal health as determined by personal medical history, clinical examination and laboratory examinations within the clinically acceptable reference range.
* Subjects having clinically acceptable 12-lead electrocardiogram (ECG).
* Subjects having clinically acceptable chest X-Ray (PIA view).
* Subjects having negative urine screen for drugs of abuse (including amphetamines, barbiturates, benzodiazepines, marijuana, cocaine, and morphine).
* Subjects having negative alcohol breath test.
* Subjects willing to adhere to the protocol requirements and to provide written informed consent.

Exclusion Criteria:

The subjects were excluded from the study, if they meet any of the following criteria:

* Hypersensitivity to Mycophenolate Mofetil or related drugs.
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder.
* History or presence of significant alcoholism or drug abuse in the past one year.
* History or presence of significant smoking (more than 10 cigarettes day or consumption of tobacco products).
* History or presence of asthma, urticaria or other significant allergic reactions.
* History or presence of significant gastric and/or duodenal ulceration.
* History or presence of glaucoma, prostatic hypertrophy or obstruction of the bladder neck, cardio-spasm and myasthenia gravis.
* History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumor.
* History or presence of cancer.
* Difficulty with donating blood.
* Difficulty in swallowing solids like tablets or capsules.
* Use of any prescribed medication or OTC medicinal products during the last two week prior to initiation of study.
* Major illness during 3 months before screening.
* Participation in a drug research study within past 3 months.
* Donation of blood in the past 3 months before screening.
* Positive screening test for any one or more: HIV, Hepatitis B and Hepatitis C.
* History or presence of significant easy bruising or bleeding.
* History or presence of significant recent trauma.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2009-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | Pre-dose, 0.083, 0.167, 0.25, 0.333, 0.41, 0.50, 0.667, 0.833, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00, 60.00 and 72.00 post dose

CONTACTS AND LOCATIONS:
Overall Officials: Jinesh Shah, MD, Principal Investigator — veeda clinical research Pvt. Ltd
Locations (1):
- veeda clinical research Pvt. Ltd, Ahmedabad, Gujarat, India